CLINICAL TRIAL: NCT07214909
Title: Gastric Emptying for Liquids of Different Volumes In Adults
Brief Title: Gastric POCUS Clear Liquids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Robert Jones, Emergency Medicine Physician, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00000214
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Gastric Emptying Time
Keywords: Gastric emptying time

STUDY DESIGN:
Intervention Model Description: Once eligibility was established, participants were randomly divided into 2 groups: one group assigned to drink 16 ounces of cold black coffee without creamer and the other group assigned to drink 16 ounces of cold black coffee with two standard creamer pods (0.76 oz) added. Randomization was generated by alternating participants between receiving black coffee or coffee with creamer after they had been consented for the study.
Who Masked: Investigator
Masking Description: Individual performing the gastric ultrasound was blinded as to which arm the study participants were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffee (Active Comparator): Study participants ingested black coffee
  Interventions: Other: Ingesting coffee without creamer
- Coffee with creamer (Experimental): Study participants ingested coffee with creamer
  Interventions: Other: Ingesting coffee with creamer

INTERVENTIONS:
Other: Ingesting coffee without creamer — Ingesting coffee without creamer and evaluating gastric emptying with gastric ultrasound at different time points.
  Arms: Coffee
Other: Ingesting coffee with creamer — Ingesting coffee with creamer and evaluating gastric emptying with gastric ultrasound at different time points.
  Arms: Coffee with creamer

SUMMARY:
To determine the gastric emptying time for clear liquids at different volumes in the adult population, for use in determining anesthesia guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Able to provide informed consent and verbally disclose their medical history in English. The study staff will not be accessing the subjects electronic medical record to verify the criteria.

Exclusion Criteria:

* Daily medications excluding oral contraceptives
* Medical conditions affecting gastric emptying, including diabetes, known gastric condition, prior gastric surgery, or pregnancy
* Inability to tolerate 7 hours of fasting
* Non-empty gastric antrum on baseline ultrasound

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Gastric emptying times of liquids at set volumes. | Study participants have a baseline ultrasound to confirm if stomach was empty and then have scans every hour after ingesting coffee until stomach was empty (Grade 0) or 4 hours maximum, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealthMC, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No